CLINICAL TRIAL: NCT00184080
Title: A Multicenter Open-Label Non-Randomized Phase II Study of Elsamitrucin (SPP 28090) in Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Brief Title: Elsamitrucin (SPP 28090) in Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Luigi Lenaz, Spectrum Pharmaceuticals, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13NHL-04-1
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

INTERVENTIONS:
Drug: Elsamitrusin

SUMMARY:
The purpose of this study is to evaluate the safety of an experimental drug called Elsamitrucin in people with non-Hodgkin's lymphoma and to see if it can shrink their tumors. Elsamitrucin has not been approved by the Food and Drug Administration (FDA). However, the FDA is permitting the use of this drug for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NHL both B and T-cell that is refractory to or has relapsed after standard therapy or for which there is no known effective treatment.
* CT or MRI scans confirming measurable tumor size (lymph node must be >1.0 cm in its longest transverse diameter). Measurement by PE is acceptable, in the case of palpable and reproducibly measurable tumors. Patients with CLL/smal lymphocytic lymphoma are eligible without bidimensional measurable disease.
* ECOG Performance Status 0-2
* Age greater or equal to 18 years of old
* AGC greater or equal to 1.0; platelets greater or equal to 75,000;Ggb greater or equal to 9.0. (Lower values may be accepted for cytopenias due to bone marrow involvement by lymphoma, after discussion with sponsor)
* Bilirubin less or equal to 2.0; SGOT and SGPT less of equal to 3 times upper limit of normal
* Creatinine <1.5; BUN <25
* Expected survival >6 months

Exclusion Criteria:

* Prior therapy with Elsamitrucin
* Any therapy for lymphoma, including chemotherapy, antibody therapy, RT, or any investigational therapy within 28 days prior to study drug administration
* Steroid therapy within the last 4 weeks prior to study drug administration
* Evidence of clinically significant uncontrolled condition/s and/or is considered by investigator to be unable to tolerate the required therapy or procedures
* Known AIDS syndrome or HIV-associated complex (severely depressed immune system)
* Prior or other current malignancy within 5 years, except for adequately treated cone-biopsied in-situ cervical cancer or resected basal cell or squamous cell skin cancer
* Any current medical or psychiatric disease that would prevent informed consent and expected cooperation of the patient for therapy and follow-up
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2004-05; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Mohrbacher, MD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States